CLINICAL TRIAL: NCT02892877
Title: The French National Reference Centre of Gestational Trophoblastic Disease
Brief Title: The French National Reference Centre of GTD
Acronym: French GTDC
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0519
Record Dates: First submitted 2016-08-02; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-08

CONDITIONS: Neoplasm, Trophoblastic; Gestational Trophoblastic Disease; Hydatidiform Mole; Hydatidiform Mole, Invasive
Keywords: Complete Hydatidiform mole; Partial Hydatidiform mole; Invasive mole; Choriocarcinoma; Post-molar neoplasia; Placental Site Trophoblastic Tumor (PSTT); Epithelioid Trophoblastic Tumor (ETT); hCG follow-up
MeSH Terms: conditions — Trophoblastic Neoplasms; Gestational Trophoblastic Disease; Hydatidiform Mole; Hydatidiform Mole, Invasive; Choriocarcinoma; Trophoblastic Tumor, Placental Site

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Complete Hydatidiform mole and Partial Hydatidiform mole
- Invasive mole
- Choriocarcinoma
- Post-molar neoplasia
- Placental Site Trophoblastic and Epithelioid Tumor

SUMMARY:
The French Gestational Trophoblastic Disease (GTD) centre has been set up and active by registering, monitoring and treating women with GTD since november 1999. The aim is to improve the management of trophoblastic disease in France.

About 850 new cases are registered each year and 140 women treated, mostly with chemotherapy and surgery.

The center works as follow, based on a multidisciplinary approach. The policy is that patient remains followed by her local physician, but can be seen and treated in the Center at demand and that the registry is done on a voluntary basis.

Each administrative french area has a local expert team (oncologist and gynaecologist) who is able to look after the patients with the help of the national reference center physicians based in Lyon.

* Once a doctor discovers a molar pregnancy, he contacts the center, with the agreement of his patient, for an opinion, an advice or simply to report the case.
* The center sends to the doctor the informed consent form to be signed by the patient, a registering form and information about pathology for patient and physician, and first guidelines based on initial pathology report.

The patient remains followed by her gynecologist, who stays her first interlocutor throughout the whole process and she goes to her local laboratory for hCG monitoring;

* A letter is sent to the initial pathology laboratory that originally carried the diagnosis of molar pregnancy to require slide sending to the pathologist referral center (9 experts with a specific pathologist national network) that centrally review initial diagnosis.
* In the mean time, the data manager collects weekly hCG values to establish a follow-up chart. The physician is regularly informed by mail of the hCG evolution.
* The local physician is contacted in case of modification of the diagnosis by the pathologist expert. The center informs him about length and monitoring methodology.
* Emails or letters are sent at each step of the management (at inclusion, at hCG negativation, and at the end of hCG follow-up).
* In case of abnormal hCG evolution (raise, plateauing or positivity at 6 months,) or if a neoplasia is anatomopathologically diagnosed (choriocarcinoma, PSTT or ETT), physician is immediately contacted by phone or email by referent gynaecologist. A complete work up including pelvic US with Doppler, pelvic MRI, thoraco-abdominal CT-scan with chest radiography if pulmonary nodules are present and brain MRI, is planned to determine the adequate treatment.

Very briefly, based on imaging results, FIGO stade and score are calculated to determine the risk. In case of low-risk, a monochemotherapy is settled, while a polychemotherapy is started in case of high-risk disease.

The investigators have developped specific expertise at key levels of diagnosis, management, follow-up, fertility preservation and treatment.

Assignments :

* Registration and monitoring post diagnosis of complete or partial molar pregnancy, choriocarcinoma,PSTT, ETT, atypical placental site nodules
* Histopathological analysis and genetics services
* Measurement of human chorionic gonadotrophin (hCG) isoforms
* Complex gynaecological surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they have a histologically proven trophoblastic disease, or a diagnosis of gestational trophoblastic neoplasia done on an abnormal evolution of hCG

Exclusion Criteria:

* none

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient diagnosed with trophoblastic disease
Sampling Method: Non-Probability Sample
Enrollment: 25500 (Estimated)
Dates: Start 1999-11; Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Agreement (yes or no) between local and pathologists in case of diagnosis of trophoblastic deseases | 18 months
  trophoblastic deseases can be partial or complete molal pregnancy, choriocarcinoma, , placental site trophoblastic tumors (PSTT), epithelioid trophoblastic tumors (ETT), atypical placental site nodule.

CONTACTS AND LOCATIONS:
Overall Officials: François Golfier, Pr, Principal Investigator — Centre National de Référence des maladies trophoblastiques Centre Hospitalier Lyon Sud - Hospices Civils de Lyon
Locations (1):
- Centre des Maladies Trophoblastiques Centre Hospitalier Lyon Sud-Bâtiment 3B-2ème étage, 165 Chemin du Grand Revoyet, Pierre-Bénite, France

REFERENCES:
- See also: Related Info — http://www.mole-chorio.com